CLINICAL TRIAL: NCT05230992
Title: Optimization of the Sensitivity of Histological Diagnosis of Pulmonary Nodules Using Cryoprobes Versus Standard Biopsy Forceps During Distal Sampling Guided by Mini Radial Ultrasound Probes
Brief Title: Optimization of the Sensitivity of Histological Diagnosis of Pulmonary Nodules
Acronym: CRYOPROBE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elsan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CRYOPROBE; 2021-A01209-32 (Other: ANSM)
Record Dates: First submitted 2021-09-24; First posted 2022-02-09 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Nodule

STUDY DESIGN:
Intervention Model Description: This is a clinical investigation of a CE (Communauté Européenne)-marked medical device that is monocentric, interventional, prospective, comparative, randomized, open-label, with cross-over design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryoprobes First (Experimental): Use of cryoprobes and then conventional forceps during the same operating time.
  Interventions: Device: Cryoprobes First
- Cryoprobes Second (Experimental): Use of conventional forceps and then cryoprobes during the same operating time.
  Interventions: Device: Cryoprobes Second

INTERVENTIONS:
Device: Cryoprobes First — In this experimental group, the Cryoprobe is used in first and the classic biopsy forceps in a second time. This medical device under study is the flexible, single-use Cryoprobe, supplied in sterile condition, 1.1 mm in diameter, 1150 mm long, with extraction tube, 817 mm long (reference 20402-401), or 757 mm long (reference 20402-402) marketed. These cryoprobes are covered by a CE marking. Cryoprobes must be used in conjunction with the Erbecryo®2 device and its accessories.
  Arms: Cryoprobes First
Device: Cryoprobes Second — In this second experimental group, the same medical devices are used but in the other order.
  Arms: Cryoprobes Second

SUMMARY:
In pulmonary oncology, the diagnosis of medium-sized pulmonary nodules (10 to 20 mm), too distal to be reached by standard bronchial fibroscopy but remaining proximal, is difficult.

There are 2 techniques: transthoracic puncture-biopsy under CT scan, usually performed by radiologists, and distal sampling guided by radial ultrasound mini-probe.

The limitations of the last technique could be overcome by the use of cryoprobes for sampling, as they would take more tissue by freezing.

DETAILED DESCRIPTION:
Concerning the interventional pneumology technique, it is performed in two steps: identification of the mass with the mini ultrasound probe and then distal sampling with a small biopsy forceps. Experience shows that there is a significant difference between the identification of the mass, which is fairly conclusive, and the samples, which are much less productive (60% at best), because it is necessary that :

* that the tumor is endo-bronchial,
* that the forceps open sufficiently to take samples by back and forth movements
* but, on the other hand, that the bronchus is not too wide.

The use of cryoprobes would allow to take more tissue by freezing. The target tissue freezes at the tip of the cryoprobe and can be detached by traction. The longer the freezing time, the more tissue is removed.

Various studies of endo-bronchial visible tumor diagnosis have compared these 2 sampling techniques (cryoprobe and conventional biopsy forceps). The cryoextraction technique performed by cryoprobes has a superior diagnostic yield (compared to flexible forceps biopsy) due to large biopsies and superior quality of the biopsied tissue (very few crush artifacts or hematomas; the morphological structure remains intact).

In this context, it seems interesting to compare these 2 techniques but in distal situation, under ultrasound detection with the mini-probes, for tumors not visible in endo-bronchial. The first samples taken in the investigating center by this technique are convincing.

In the framework of this study, in the same operating time and after ultrasound identification of the tumor, biopsies will be performed by conventional forceps (5 samples) and by cryoprobes (3 samples) on the same site. The sequence of use of one or the other technique will be randomly selected. Thus, each patient is his own control.

This first pilot study will explore the feasibility, effectiveness and safety of this procedure. Depending on the results of this comparative study, a second study including more patients will validate this procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a tumor of any location with a draining bronchus (primary lung cancer or lung metastases)
* Suspected lung nodule(s) with anatomical situation on mid 1/3 CT
* Presence of at least one lung nodule of sufficient size on CT to allow for at least 8 tissue samples
* Male or female aged ≥ 18 years
* Mandatory membership in a health insurance plan
* Patient who has been informed about the study and has signed the informed consent form

Exclusion Criteria:

* Proximal or distal pulmonary nodule(s)
* Pacemaker patient
* Pregnant or nursing women
* Patients under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-11-05 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Validity of samples by cryoprobes | Within 24 hours after intervention
  Histological diagnosis from the material collected by cryoprobes and conventional forceps

SECONDARY OUTCOMES:
Specificity, sensitivity, and predictive values of each technique | Within 24 hours after intervention
  specificity, sensitivity, predictive values
Tolerance and safety of the samples taken | 15 Days after intervention
  Collection of adverse events for the duration of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Pneumologie Elsan Santé Atlantique, Saint-Herblain, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dhooria S, Sehgal IS, Aggarwal AN, Behera D, Agarwal R. Diagnostic Yield and Safety of Cryoprobe Transbronchial Lung Biopsy in Diffuse Parenchymal Lung Diseases: Systematic Review and Meta-Analysis. Respir Care. 2016 May;61(5):700-12. doi: 10.4187/respcare.04488. Epub 2016 Mar 1. PMID 26932382
- [Background] Hagmeyer L, Theegarten D, Treml M, Priegnitz C, Randerath W. Validation of transbronchial cryobiopsy in interstitial lung disease - interim analysis of a prospective trial and critical review of the literature. Sarcoidosis Vasc Diffuse Lung Dis. 2016 Mar 29;33(1):2-9. PMID 27055830
- [Background] Montufar F, Moral LD, Labarca G, Folch E, Majid A, Fernandez-Bussy S. [Transbronchial cryobiopsies and cryotherapy in lung diseases]. Rev Med Chil. 2018 Sep;146(9):1033-1040. doi: 10.4067/s0034-98872018000901033. Spanish. PMID 30725025
- [Background] Gershman E, Fruchter O, Benjamin F, Nader AR, Rosengarten D, Rusanov V, Fridel L, Kramer MR. Safety of Cryo-Transbronchial Biopsy in Diffuse Lung Diseases: Analysis of Three Hundred Cases. Respiration. 2015;90(1):40-6. doi: 10.1159/000381921. Epub 2015 May 20. PMID 25998966
- [Background] Schumann C, Hetzel J, Babiak AJ, Merk T, Wibmer T, Moller P, Lepper PM, Hetzel M. Cryoprobe biopsy increases the diagnostic yield in endobronchial tumor lesions. J Thorac Cardiovasc Surg. 2010 Aug;140(2):417-21. doi: 10.1016/j.jtcvs.2009.12.028. Epub 2010 Mar 11. PMID 20226474
- [Background] Hetzel J, Eberhardt R, Herth FJ, Petermann C, Reichle G, Freitag L, Dobbertin I, Franke KJ, Stanzel F, Beyer T, Moller P, Fritz P, Ott G, Schnabel PA, Kastendieck H, Lang W, Morresi-Hauf AT, Szyrach MN, Muche R, Shah PL, Babiak A, Hetzel M. Cryobiopsy increases the diagnostic yield of endobronchial biopsy: a multicentre trial. Eur Respir J. 2012 Mar;39(3):685-90. doi: 10.1183/09031936.00033011. Epub 2011 Aug 18. PMID 21852332